CLINICAL TRIAL: NCT04581746
Title: Evaluation of the Impact of the Epidemic of COVID-19 Infection Among People Living With HIV (SARS-CoV-2)
Brief Title: Impact of the Epidemic of COVID-19 Infection Among People Living With HIV (SARS-CoV-2)
Acronym: coVIHd-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIPH_2020_7
Record Dates: First submitted 2020-09-22; First posted 2020-10-09 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Virus-HIV; Covid19
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Other): questionnaire and follow-up visit
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — bi-monthly questionnaire and then one visit with questionnaire and covid-19 test

SUMMARY:
The non-essential and non-urgent follow-up consultations of patients living with HIV were postponed or transformed into "teleconsultation" or exchanges of e-mails between practitioners and patients during COVID-19 epidemic. This change in care can have an impact on follow-up and access to treatment for PVVIH.

DETAILED DESCRIPTION:
On 16 March 2020, an instruction to postpone "non-urgent" consultations was given to doctors. Thus, the non-essential and non-urgent follow-up consultations of patients living with HIV were postponed or transformed into "teleconsultation" or exchanges of e-mails between practitioners and patients. This change in care can have an impact on follow-up and access to treatment for PVVIH. In addition, the epidemic itself may have consequences: PVVIH may be at greater risk because of their immunosuppression and associated co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed up for HIV infection in one of the COREVIH Hauts de France centres participating in the study
* Having communicated an email address
* Having given their consent to participate in this study
* Beneficiary subject affiliated or entitled to a social security scheme

Exclusion Criteria:

* Minor patient
* Refusal to participate
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SARS CoV2 infection in PVVIH in Hauts de France | Inclusion
  Determination of the number of patients with microbiologically or clinically-biologically proven SARS CoV2 infection at inclusion in the study

SECONDARY OUTCOMES:
Prevalence of SARS CoV2 infection in PVVIH in Hauts de France | through study completion, an average of 19 months
  Determination of the number of patients with microbiologically or clinically-biologically proven SARS CoV2 infection at the end of the study
Determine the incidence rate of COVID 19 among PVVIH antiretroviral treatment | through study completion, an average of 19 months
  Percentage of patients who stopped their antiretroviral treatment
Determine the incidence rate of COVID 19 among PVVIH discontinuing antiretroviral treatment | through study completion, an average of 19 months
  Reason for discontinuing antiretroviral treatment
Determine the incidence rate of COVID 19 among PVVIH who stopped all follow-up | through study completion, an average of 19 months
  Percentage of patients who stopped all follow-up by an infectious disease specialist
Psychological consequences of this epidemic among PVVIH : HAD | through study completion, an average of 19 months
  Evaluation of the psychological scales HAD on PVVIH
Psychological consequences of this epidemic among PVVIH : PROQOL-HIV | through study completion, an average of 19 months
  Evaluation of the psychological scales PROQOL-HIV on PVVIH

CONTACTS AND LOCATIONS:
Overall Officials: Pauline THILL, MD, Principal Investigator — CH TOURCOING
Locations (3):
- France (3):
  - CHU Amiens Picardie, Amiens
  - CH Lens, Lens
  - CH Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: No